CLINICAL TRIAL: NCT04062955
Title: Adherence to the Alternative Healthy Eating Index and Effects on Inflammatory Markers and Breast Density
Brief Title: Effects of Alternative Healthy Eating Index-Based Diet on Inflammatory Markers and Breast Density in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1001812; NCI-2019-05132 (Registry Identifier: NCI / CTRP); 8665 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-08-13; First posted 2019-08-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Healthy Subject
Keywords: Breast - Female
MeSH Terms: interventions — Diet Therapy; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (dietary intervention) (Experimental): DIETARY INTERVENTION: Participants receive dietary counseling with a dietitian in person or via telephone to support adherence to a diet based on the AHEI guidelines once weekly for up to 12 weeks.
  DXA ONLY STUDY: Participants undergo DXA scan for breast density measurement at baseline and at 12 weeks.
  Interventions: Dietary Supplement: Dietary Intervention; Procedure: Dual X-ray Absorptiometry; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Receive dietary counseling
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Procedure: Dual X-ray Absorptiometry — Undergo DXA scan
  Other Names: BMD scan; bone mineral density scan; DEXA; DEXA Scan; dual energy x-ray absorptiometric scan; Dual Energy X-ray Absorptiometry; Dual X-Ray Absorptometry; DXA; DXA SCAN
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the effects of a dietary intervention based on the Alternative Healthy Eating Index (AHEI) on inflammatory markers and breast density in healthy participants. The AHEI is a quantifiable measure of diet quality designed to target food and macronutrient sources that are associated with chronic disease risk. Adherence to the AHEI may be associated with a reduction in inflammatory biomarkers and sex steroid hormone levels compared to other dietary patterns/scores.

DETAILED DESCRIPTION:
OUTLINE:

DIETARY INTERVENTION: Participants receive dietary counseling with a dietitian in person or via telephone to support adherence to a diet based on the AHEI guidelines once weekly for up to 12 weeks.

DUAL X-RAY ABSORPTIOMETRY (DXA) ONLY STUDY: Participants undergo DXA scan for breast density measurement at baseline and at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women will be eligible if they are nulliparous, aged 18-30, and score below 75 on the AHEI. Study eligibility will be assessed via online screening questionnaire and online Food Frequency Questionnaire (FFQ). These criteria were chosen because of our focus on the years before first birth as a critical period for establishing breast cancer risk
* Participants must be able to come to two clinic visits, complete questionnaires in English, and will be required to discontinue all vitamins and nutritional supplements during the study period
* DXA ONLY PILOT STUDY: Participants must be able to come to one visit in the Prevention Center where they will receive the consent form and undergo the DXA scan. No intervention will occur and there will be no follow-up assessments or measurements beyond the DXA scan

Exclusion Criteria:

* Women will be ineligible if they are postmenopausal, pregnant, taking hormone therapy (e.g., oral contraceptives), or have chronic illnesses that are known to affect gastrointestinal absorption of nutrients
* Women who obtain a score of >= 75 on the AHEI are also ineligible
* DXA ONLY PILOT STUDY: Women who are pregnant

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory markers (IL-6, IL-1β, CRP, sTNFR-1, sTNFR-2, hsCRP) | At baseline and week 12
  Levels of IL-6, IL-1β, sTNFR-1, and sTNFR-2 will be measured by immunoassay. hsCRP levels will be measured using a high-sensitivity latex-enhanced immunonephelometric assay on a BNII analyzer.
Change in breast density | At baseline and week 12
  Breast density will be measured by dual x-ray absorptiometry. Depending on the distribution of the data a paired t-test or Wilcoxon signed-rank test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Harris, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No